CLINICAL TRIAL: NCT00566410
Title: A Phase I, Open-Labeled, Single-Arm, Dose Escalation, Clinical and Pharmacology Study of Dichloroacetate (DCA) in Patients With Recurrent and/or Metastatic Solid Tumours
Acronym: DCA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AHS Cancer Control Alberta (Other)
Collaborators: Cross Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23596; NCT00570076 (obsolete NCT alias)
Record Dates: First submitted 2007-11-29; First posted 2007-12-03 (Estimated); Last update posted 2016-03-11 (Estimated); Status verified 2016-03

CONDITIONS: Neoplasms
Keywords: DCA; Phase I; Dose Escalation; Solid Tumours; Dichloroacetate; Pharmacokinetic
MeSH Terms: conditions — Neoplasms | interventions — Dichloroacetic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Dichloroacetate — Continuous daily oral dosage (bid).

SUMMARY:
Dichloroacetate (DCA) is a small molecule that has been used for years to treat lactic acidosis and rare metabolic disorders in humans. Further testing now shows that it may suppress the growth of human cancer cells. Tests of DCA on human cells cultured outside of the body found that it killed lung, breast, and brain cancer cells, without affecting human normal cells. Tumors in rats that were infected with human tumors also shrank considerably. Most cancers are characterized by a resistance to apoptosis (cell death that removes abnormal cells) that makes them more likely to grow as well as be resistant to most cancer treatments. Plus, many current cancer treatments kill both cancerous and healthy cells and are highly toxic. DCA works by reversing the damage to the mitochondria that is present in cancer cells, thus reactivating the apoptosis (cell death) mechanism in them. The result is the death of the cancer cells. This mitochondrial reactivation presents an entirely new approach to treating cancer.

DCA is known to be relatively well tolerated with few significant side effects and its selectivity, effectiveness and ease of delivery (oral) make it an attractive opportunity. It is hoped that one day this treatment may become a safe and effective treatment, either along or in conjunction with other treatments, for many forms of cancer.

DETAILED DESCRIPTION:
As cancer cells have a hyperpolarized mitochondrial membrane and deficiency in Kv channel expression, it was postulated that the reversal of this observation may increase apoptosis and inhibit tumor growth. Bonnet and colleagues reported that the administration of DCA led to the switch from glycolysis to oxidative phosphorylation in the Krebs Cycle through inhibition of PDHK. This was associated with an increase in the production of reactive oxygen species and a decrease in hyperpolarization of the inner mitochondrial membrane, leading to efflux of proapoptotic proteins and apoptosis as measured by increased in TUNEL-positive cells. In addition, DCA also decreased the expression of survivin, an anti-apoptotic protein. DCA upregulated the expression of Kv channels in cancer cells, leading to efflux of potassium ions and further increased the proapoptotic effect of DCA. Such change in energy metabolism and apoptosis was not observed in normal cells. DCA was also shown to inhibit tumor growth both in vitro and in vivo. Thus, inhibition of PDHK by DCA represents a novel anti-cancer therapy target with reasonable toxicities to normal tissue. It is therefore of interest to study DCA in refractory cancer patients.

Although the bioavailability was only 50-60% in normal subjects treated with 2.5 microgram/kg of DCA , in a study using clinically relevant dose of DCA at 50 mg/kg, the bioavailability was 100% in health volunteers. DCA administered at 50 mg/kg/day can achieve plasma concentrations above those require for inhibition of PHDK, the target enzyme for at least 24 hours, without exceeding the concentration for maximal lactate lowering. There was a high incidence of peripheral neuropathy in adults with MELAS after administration of DCA at 50 mg/kg/day for 6 months, but peripheral neuropathy is part of the MELAS syndrome, and many adult patients with MELAS develop diabetes mellitus, which commonly presents with peripheral neuropathy. In the contrary, no peripheral neuropathy was observed in children with congenital acidosis after prolonged treatment with DCA at 50 mg/kg/day up to 2 years. Therefore, with exclusion of patients with any grade 2 or higher peripheral neuropathy and with careful monitoring of peripheral neuropathy using monofilaments, the likelihood of developing severe peripheral neuropathy in adult cancer patients should be minimized. Given the presence of significant neuropathy in adult patients with MELAS after treatment with DCA at 25 mg/kg/day, it is judged to be safe and reasonable to establish the starting dose at 12.5 mg/kg/day in adult cancer patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologically or cytologically confirmed recurrent or metastatic solid tumours. All patients will have no meaningful therapies available to them including hormone therapy, chemotherapy and targeted therapies. For the malignancies that have no proven therapy, they can be enrolled without any prior systemic therapy.
2. Four weeks must have elapsed since prior chemotherapy, hormonal therapy, targeted therapy, or radiation therapy. There is no restriction in the amount of bone marrow previously radiated.
3. Recovery to baseline or, at most, grade 1 of all drug-related toxicities due to prior chemotherapy, radiation, hormonal therapy, or molecular targeted therapy, except for alopecia.
4. Age ≥ 18 years.
5. ECOG performance status ≤ 2 (Karnofsky ≥70%, see Appendix A).
6. Life expectancy of greater than 12 weeks.
7. Patients must have normal organ and marrow function as defined below:

   * absolute neutrophil count ≥1,500/mcL
   * hemoglobin ≥90 g/L
   * platelets ≥100,000/mcL
   * total bilirubin ≤1.5 X upper limit of normal (ULN)
   * AST(SGOT) and ALT(SGPT) ≤2.5 X ULN or ≤ 5 X ULN in the presence of liver metastases
   * creatinine ≤1.5 X institutional upper limit of normal
8. Cardiac ejection fraction by MUGA scan or echocardiogram must be >50% for patients at baseline.
9. The effects of DCA on the developing human fetus are unknown. For this reason and because DCA can be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (e.g.: hormonal or barrier method of birth control, abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
10. Ability to understand the purpose of the study and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Patients who have had chemotherapy, hormonal therapy, molecular targeted therapy, or radiotherapy within 4 weeks prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier.
2. Patients may not be receiving any other investigational agents, chemotherapy, immunotherapy, radiotherapy, or molecular targeted agents.
3. Patients with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that could confound the evaluation of neurologic and other adverse events.
4. History of allergic reactions attributed to compounds of similar chemical or biologic composition to DCA.
5. Due to the possibility of peripheral sensorimotor neuropathy from DCA, the presence of grade 2 or higher peripheral neuropathy due to prior medical condition (such as multiple sclerosis), medications, or other etiologies.
6. Any psychological, familial, sociological, or geographical conditions that do not permit medical follow-up and compliance with the study protocol.
7. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements. Specifically, for patients who are taking either or both oral hypoglycemics and insulin for diabetes mellitus will not be eligible as DCA in combination with these agents may increase the risk of clinically significant hypoglycemia, compromising patient safety.
8. Pregnant women are excluded from this study because DCA is an agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with DCA, breastfeeding should be discontinued if the mother is treated with DCA.
9. HIV-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with DCA. In addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy. Appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated.
10. 5 years must have elapsed since the initial curative procedure for other malignancies, except for in situ cervical cancer, basal cell carcinoma of the skin, and localized prostate cancer after curative therapy such as surgery, or radiation.
11. History of malabsorption syndrome or substantial amount of small bowels or stomach removed that may impair absorption of DCA.
12. Patients taking warfarin. Low dose or therapeutic dose of heparin or low molecular weight heparin is allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2007-12; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
To assess safety and tolerability of oral DCA | Trial Completion
To determine the dose-limiting toxicity (DLT) and phase II dose | Trial completion
To characterize pharmacokinetic (PK) profile | Trial Completion

SECONDARY OUTCOMES:
To evaluate the effect of oral DCA | Trial Completion
To evaluate the clinical response rate | Trial completion
To evaluate the change in standard uptake value by FDG-PET scans before and after treatment with DCA | Trial completion

CONTACTS AND LOCATIONS:
Overall Officials: Peter Venner, M.D., Principal Investigator — AHS Cancer Control Alberta; Evangelos Michelakis, M.D., Principal Investigator — University of Alberta
Locations (1):
- Cross Cancer Institute, Edmonton, Alberta, Canada